CLINICAL TRIAL: NCT02507336
Title: Long-term Follow-up and/or Continued Thalidomide (THALOMID®) Maintenance Therapy for Patients Enrolled on Clinical Trial 20030165
Brief Title: Long-Term Followup and/or Thalidomide Maintenance Therapy for Patients Enrolled on Clinical Trial 20030165
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Izidore Lossos, MD, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20150402
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Mantle Cell Lymphoma; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A - CR+Thalidomide (Experimental): Patients who achieved complete response (CR) in 20030165 and continue to receive maintenance Thalidomide. Patients in Group A will receive daily oral thalidomide (THALOMID®) as per standard of care and THALOMID® REMS™ guidelines. Patients will continue with thalidomide (THALOMID®) as per standard of care guidelines, until progression of disease, discontinuation due to toxicity, death or study withdrawal. Patients will receive annual clinical/laboratory evaluations.
  Interventions: Drug: Thalidomide
- Group B - CR+No Thalidomide (No Intervention): Patients who achieved complete response (CR) in 20030165, but are not receiving maintenance Thalidomide. Patients will receive annual clinical/laboratory evaluations.
- Group C - PD or Expired (No Intervention): All other patients enrolled in 20030165 who expired or experienced disease progression (PD). Patients will be followed annually for survival.

INTERVENTIONS:
Drug: Thalidomide — 100-300 mg capsule taken by mouth once daily.
  Other Names: Thalomid
  Arms: Group A - CR+Thalidomide

SUMMARY:
The study seeks to provide long-term follow-up and/or to offer continued maintenance thalidomide (THALOMID) therapy to those patients enrolled in 20030165. Patients will be followed until withdrawal of consent, or death.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled on the 20030165 clinical trial.
2. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who were discontinued from 20030165 for any reason prior to the completion of protocol-specified treatment (e.g. withdrawal of consent).
2. Uncontrolled, intercurrent serious illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, and/or cardiac arrhythmia likely in the judgment of the PI to interfere with clinical study requirements.
3. Psychiatric illness/condition likely in the judgment of the PI to limit compliance with clinical study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Izidore Lossos, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lossos IS, Hosein PJ, Morgensztern D, Coleman F, Escalon MP, Byrne GE Jr, Rosenblatt JD, Walker GR. High rate and prolonged duration of complete remissions induced by rituximab, methotrexate, doxorubicin, cyclophosphamide, vincristine, ifosfamide, etoposide, cytarabine, and thalidomide (R-MACLO-IVAM-T), a modification of the National Cancer Institute 89-C-41 regimen, in patients with newly diagnosed mantle cell lymphoma. Leuk Lymphoma. 2010 Mar;51(3):406-14. doi: 10.3109/10428190903518345. PMID 20038221

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A - CR+Thalidomide
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group A - CR+Thalidomide
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the length of time, during and after treatment, until documented disease progression or death (by any cause, in the absence of progression).
Time Frame: Up to five years
Measure: Number; unit: years
Arm/Group | Group A - CR+Thalidomide
Number analyzed (Participants) | 2
years | NA — Results not reported due to participant confidentiality.

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the elapsed time from start of treatment until death or date of censoring.
Time Frame: Up to five years
Population: Results not reported due to participant confidentiality.
Measure: Number; unit: years
Arm/Group | Group A - CR+Thalidomide
Number analyzed (Participants) | 2
years | NA — Results not reported due to participant confidentiality.

3. Secondary Outcome: Response Rate (RR)
Description: Response rate is defined as the percentage of participants whose cancer shrinks or disappears after treatment.
Time Frame: Up to five years
Measure: Number; unit: percentage of participants
Arm/Group | Group A - CR+Thalidomide
Number analyzed (Participants) | 2
percentage of participants | NA — Results not reported due to participant confidentiality.

4. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Description: Treatment emergent adverse events will be assessed by treating physician using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 3.0.
Time Frame: Up to five years
Measure: Number; unit: percentage of participants
Arm/Group | Group A - CR+Thalidomide
Number analyzed (Participants) | 2
percentage of participants | NA — Results not reported due to participant confidentiality.

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Adverse Events not reported due to participant confidentiality.
Arm/Group | Group A - CR+Thalidomide
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
To protect participant privacy and maintain confidentiality, results will not be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT02507336/Prot_000.pdf